CLINICAL TRIAL: NCT03669341
Title: Short-term Apnoea Training With Deep Inspiration Breath Hold vs High Frequency Percussive Ventilation for Apnoea-like Suppression of Respiratory Motion: a Pilot Study Using Magnetic Resonance Imaging at 1.5T Assessing Their Application for Proton Therapy Treatment of Lung Tumors
Brief Title: Assessment of 2 Different Techniques for Suppression of Respiratory Motion in Lung Cancer Treatment With Proton Therapy Using Magnetic Resonance Imaging (MRI)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Paul Scherrer Institut, Center for Proton Therapy (Other)
Collaborators: Swiss Federal Institute of Technology (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: APNOPART_2018
Record Dates: First submitted 2018-09-11; First posted 2018-09-13 (Actual); Last update posted 2021-06-09 (Actual); Status verified 2021-06

CONDITIONS: Healthy Volunteers
Keywords: breath hold; DIBH; HFPV; MRI

STUDY DESIGN:
Intervention Model Description: All study participants will perform both techniques of suppression of respiratory motion at 4 weekly visits. They always start with the deep-inspiration-breath- hold (DIBH) technique, extended by prior hyperventilation while breathing 100% O2, followed by the high-frequency-percussive-ventilation (HFPV) technique. Inbetween the weekly visits, participants are requested to perform a daily, short breath-hold training at home.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Deep Inspiration Breath Hold (DIBH) (Experimental): DIBH extended by prior hyperventilation while breathing 100% O2
  Interventions: Other: Deep Inspiration Breath Hold (DIBH)
- High Frequency Percussive Ventilation (HFPV) (Active Comparator): passive Ventilation by a jet ventilator
  Interventions: Other: High Frequency Percussive Ventilation (HFPV)

INTERVENTIONS:
Other: Deep Inspiration Breath Hold (DIBH) — human-based DIBH method with short-term breath-hold training
  Arms: Deep Inspiration Breath Hold (DIBH)
Other: High Frequency Percussive Ventilation (HFPV) — device-based HFPV technique
  Arms: High Frequency Percussive Ventilation (HFPV)

SUMMARY:
Since 1996 proton therapy has been applied very successfully at the Paul Scherrer Institute in Switzerland to irradiate deep-seated, stationary tumors. In order to treat tumors within an organ which moves due to breathing (e.g. lung) motion mitigation strategies need to be implemented to ensure the precise irradiation of the moving target. The aim of this study is to assess the feasibility and compare (via MRI imaging) 2 techniques which "freeze" the movement of the lung by breath hold. One method is suppression of respiratory movement via high-frequency, mechanical ventilation by means of a Jet Ventilator (HFPV). The other technique is deep Inspiration breath-hold (DIBH) with Hyperventilation and simultaneous Inspiration of 100% O2 including daily breath-hold exercise.

ELIGIBILITY:
Inclusion Criteria:

* ability to give informed consent by signature
* healthy, i.e. normal physical and mental status

Exclusion Criteria:

* contraindications to MRI (non-MRI-suitable electronical & metal implants, claustrophobia)
* women who are pregnant or are breast feeding
* acute or chronic illness
* known or suspected non-compliance, drug or alcohol abuse
* inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant
* presence of any psychological or sociological condition potentially hampering compliance with the study protocol

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-10-10 (Actual); Primary Completion 2019-03-11 (Actual); Study Completion 2019-08-14 (Actual)

PRIMARY OUTCOMES:
Difference in MRI Images | 3 weeks
  pulmonary anatomical structure points are evaluated by means of MRI scans. The difference of these MRI evaluations between the DIBH- and HFPV-technique is the primary outcome measure.

SECONDARY OUTCOMES:
Difference in breath-hold duration | 3 weeks
  The difference between the DIBH- and HFPV-technique in breath-hold Duration is the secondary outcome measure

CONTACTS AND LOCATIONS:
Overall Officials: Frank Emert, PhD, Principal Investigator — Paul Scherrer Institut, Center for Proton Therapy
Locations (1):
- Paul Scherrer Institut, Center for Proton Therapy, Villigen, Canton of Aargau, Switzerland

REFERENCES:
- [Background] Emert F, Missimer J, Eichenberger PA, Walser M, Gmur C, Lomax AJ, Weber DC, Spengler CM. Enhanced Deep-Inspiration Breath Hold Superior to High-Frequency Percussive Ventilation for Respiratory Motion Mitigation: A Physiology-Driven, MRI-Guided Assessment Toward Optimized Lung Cancer Treatment With Proton Therapy. Front Oncol. 2021 Apr 29;11:621350. doi: 10.3389/fonc.2021.621350. eCollection 2021. PMID 33996545